CLINICAL TRIAL: NCT06441253
Title: Development and Evaluation of a Portable Wedge Device for Calf Stretching to Alleviate Strain and Spasms: A RCT Study
Brief Title: Development and Evaluation of a Portable Wedge Device for Calf Stretching to Alleviate Strain and Spasms
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MSRSW/Batch-Fall22/718
Record Dates: First submitted 2024-05-25; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Spasm
MeSH Terms: conditions — Spasm | interventions — Exercise Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deep Friction massage (Other)
  Interventions: Diagnostic Test: Deep Friction massage
- Therapeutic exercises (Experimental)
  Interventions: Combination Product: Therapeutic exercises

INTERVENTIONS:
Diagnostic Test: Deep Friction massage — The calf muscles received a firm, deep-circulation massage with fingertip pressure
  Arms: Deep Friction massage
Combination Product: Therapeutic exercises — Four stretching exercises were performed for twenty minutes, five minutes for each technique, and eight to ten repetitions of each exercise (calf wall stretch, back knee straight, bilateral calf stretches, knees straight, ankle plantarflexion/dorsiflexion)
  Arms: Therapeutic exercises

SUMMARY:
This research aimed to contribute valuable insights into the potential benefits of incorporating the portable wedge device into preventive or therapeutic interventions for calf-related musculoskeletal issues.

DETAILED DESCRIPTION:
By combining economical, ergonomic principles and user-friendly features, the proposed device offered individuals a convenient and efficient means to enhance their calf flexibility, ultimately mitigating strain and reducing spasms. Developing and successfully integrating a portable wedge device could mark a significant breakthrough in preventive and rehabilitative care for musculoskeletal problems associated with the calf region. This innovative device can enhance the overall well-being and musculoskeletal health of individuals suffering from such issues, providing a more effective and convenient treatment solution.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients diagnosed with Calf Strain and Spasm
* Age above 18
* Participants who are volunteer for the study
* Patients who suffer from leg pain or functional disability

Exclusion Criteria:

* Unconscious patients
* Patients with difficulty in seeing and hearing
* Patients having a history of mental illnesses (Stroke, Multiple sclerosis, Parkinsonism, Alzheimer's Disease)
* Patient history of severe mobility disorder
* Systemic illness (Liver Failure, Active cancer, Cardiopulmonary distress)
* Decline to participate in this study
* Active fracture and dislocations
* Arthritic disorders (such as osteoarthritis, Rheumatoid Arthritis, Psoriatic Arthritis, and Fibromyalgia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-10-29 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | 12 Months
  subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between 0 for "no pain" and 10 for "worst pain".
Functional Disability Scale for Ankle (FADI) | 12 months
  The FADI has 26 items. Each item is scored from 0 (unable to do) to 4 (no difficulty at all). The 4 pain items of the FADI are scored 0 (unbearable) to 4 (none). The FADI has a total point value of 104 points, whereas the FADI Sport has a total point value of 32 points.
Range of motion (ROM) | 12 months
  This tool measures the angle of dorsiflexion before and after the intervention, offering insights into the functional improvements resulting from the use of the portable wedge device. Additionally, participant satisfaction and compliance will be assessed through a structured questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Faqraj Sharif Hospital (Trust) Physiotherapy and Orthopedic Department and Ramay Clinic (Physiotherapy and Orthopedic Department), Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No